CLINICAL TRIAL: NCT03274479
Title: Phase I Trial of PBF-1129 in Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: PBF-1129 in Patients With NSCLC
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Palobiofarma SL (Industry)
Collaborators: Ohio State University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PBF-1129CT_03
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced or Metastatic NSCLC
Keywords: adenosine receptors; checkpoint inhibitors; immune system activator
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PBF-1129_40mg (Experimental)
  Interventions: Drug: PBF-1129
- PBF-1129_80mg (Experimental)
  Interventions: Drug: PBF-1129
- PBF-1129_160mg (Experimental)
  Interventions: Drug: PBF-1129
- PBF-1129_320mg (Experimental)
  Interventions: Drug: PBF-1129

INTERVENTIONS:
Drug: PBF-1129 — PBF-1129 once a day by oral administration

SUMMARY:
Phase I clinical trial in Eastern Cooperative Oncology Group (ECOG) 0-1 patients with locally advanced or metastatic NSCLC to evaluate safety and tolerability of the compound PBF-1129, an Adenosine A2b receptor antagonist. The phase I dose escalation will be conducted 3+3 method. Pharmacokinetic (PK) data will be also obtained.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological diagnosis of metastatic squamous or non-squamous NSCLC.
* Life expectancy greater or equal to 3 months, as determined by the investigator -Patients must have progressed on the standard therapy, including platinum based - chemotherapy. Patients with epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), or ROS-1 mutations must have progressed on standard treatment options including EGFR, ALK, or ROS-1-directed therapies.
* No limits to the prior lines of treatment
* ECOG performance status of 0/1
* Measurable Disease by RECIST v1.1
* Age greater than 18 years.
* Adequate bone marrow, renal and hepatic function:

  * Absolute neutrophil count (ANC) ≥ 1500 /µL
* White blood cell count (WBC) t ≥ 2.5 x 109/L (2500/µL)

  * Lymphocyte count ≥ 0.5 x 109/L (500/µL)
* Platelet count ≥ 100 x 109/L (100,000/µL) without transfusion
* Hemoglobin ≥ (9.0 g/dL) - patients may be transfused to meet this criterion.
* Aspartate aminotransferase AST, alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 2.5 x upper limit of normal (ULN)

  * Serum bilirubin ≤ 1.5 x ULN, with the exception of patients with known Gilbert disease: serum bilirubin level ≤ 3 x ULN
  * Creatinine clearance >60 mL/min (calculated using the Cockcroft-Gault formula) or by 24-hours urine collection
* Written informed consent and any locally-required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Subject is willing and able to comply with the protocol for the duration of the study

Exclusion Criteria:

* Participation in another clinical study with an investigational product during the last 4 weeks or 5 half-lives prior to starting on treatment.
* Symptomatic and/or untreated or actively progressing central nervous system (CNS) metastases or leptomeningeal disease. Patients with a history of treated CNS metastases are eligible, provided that all of the following criteria are met:

  * The patient has not received stereotactic radiotherapy within 7 days prior to initiation of study treatment or whole-brain radiotherapy within 14 days prior to initiation of study treatment.
  * The patient has no ongoing requirement for corticosteroids as therapy for CNS disease. Anti-convulsant therapy at a stable dose is permitted.
* Serious uncontrolled medical disorder or active infection that would impair the patient's ability to receive study treatment.
* Concurrent use of other anticancer approved or investigational agents is not allowed.
* Autoimmune disorder
* Prior malignancy in past 2 years or as identified in Section 7.2 of this protocol
* Active or prior documented autoimmune disease within the past 2 years. NOTE: Patients with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Patients receiving systemic steroids ≥ 10mg/day of prednisone or the equivalent
* Smoking (cigarettes, cigars or pipes) must be discontinued at least 7 days prior to initiating study drug administration; smoking cessation products (transdermal nicotine patches or chewing gum may be used.
* Pregnancy or breastfeeding, or intention of becoming pregnant during the study. Female subjects must either be of non-reproductive potential or have a negative serum pregnancy test result within 14 days prior to initiation of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of PBF-1129 | 28 days
  The MTD evaluation will be based on the Dose-limiting Toxicity (DLT) of the treated Population, which includes all subjects who receive any dose of PBF-1129, and will include Adverse events (AEs), Serious Adverse events (SAEs), laboratory evaluations and electrocardiogram (ECG) results

SECONDARY OUTCOMES:
Time to PBF-1129 peak concentration in plasma "Tmax" | days 1 and 29
  The parameter will be calculated from plasma samples collected at days 1 and 29 after drug administration.It will consist in the time (in minutes) to reach the maximum "PBF-1129" concentration in plasma samples of patients after oral administration of PBF-1129.
Time to PBF-1129 peak concentration in plasma at steady state "Tmax,ss" | days 1 and 29
  The parameter will be calculated from plasma samples collected at days 1 and 29 after drug administration.
  It will consist in the time (in minutes) to reach the maximum "PBF-1129" concentration in plasma samples of patients during a dosing interval at steady state.
PBF-1129 peak concentration in plasma "Cmax" | days 1 and 29
  The parameter will be calculated from plasma samples collected at days 1 and 29 after drug administration. It will consist in the maximum plasma concentration (ng/mL) of PBF-1129 observed after administration.
PBF-1129 peak concentration in plasma at steady state"Cmax,ss" | days 1 and 29
  The parameter will be calculated from plasma samples collected at days 1 and 29 after drug administration.It will consist in the maximum plasma concentration (ng/mL) of PBF-1129 observed during a dosing interval at steady state.
The area under PBF-1129 plasma concentration-time curve to infinite time "AUC(0-inf)" | days 1 and 29
  The parameter will be calculated from plasma samples collected at days 1 and 29 after drug administration.
  It will consist in the area under the concentration-time curve from zero up to ∞ with extrapolation of the terminal phase. "AUC(0-inf)" will be given in Amount·time/ volume units
The area under PBF-1129 plasma concentration-time curve up to time 't' "AUC(0-t)" | days 1 and 29
  The parameter will be calculated from plasma samples collected at days 1 and 29 after drug administration.It will consist in the area under the concentration-time curve from zero up to a definite time t. "AUC(0-t)" will be given in Amount·time/ volume units.
The area under PBF-1129 plasma concentration-time curve over the dosing interval "AUC(0-τ)" | days 1 and 29
  The parameter will be calculated from plasma samples collected at days 1 and 29 after drug administration. It will consist in the area under the concentration-time curve over the dosing interval. "AUC(0-τ)" will be given in Amount·time/ volume units.
PBF-1129 half-life in plasma " t½" | days 1 and 29
  The parameter will be calculated from plasma samples collected at days 1 and 29 after drug administration. It will consist in the terminal half-life of PBF-1129 in plasma. "t½" will be given in hours (h)
Efficacy as measured by Objective response rate (ORR) | 2 years
  ORR: Response and progression will be evaluated in this study using the new international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).ORR is defined as confirmed complete response (CR) or partial response (PR) based on modified RECIST v1.1.
Efficacy as measured by Disease control rate (DCR) | 2 years
  The disease control rate (DCR) will be estimated considering the following variables:
  Complete response (CR), Partial response (PR) and stable disease (SD) as described by Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1). These variables will be assessed based on Imaging-based evaluation methods as chest x-ray, conventional computed tomography (CT) and magnetic resonance imaging (MRI) that will be performed every 2 cycles of 28 days administration.
Efficacy as measured by duration of response (DoR) | 2 years
  Duration of response (DoR) is defined as the duration from the first documentation of OR to the first documented disease progression or death due to any cause, whichever occurs first
Efficacy as measured by progression-free survival (PFS) | 2 years
  Progression-free survival (PFS) will be measured from the start of treatment until the documentation of disease progression or death due to any cause, whichever occurs first. For subjects who are alive and progression-free at the time of data cut-off for analysis, PFS will be censored at the last tumor assessment date.
Efficacy as measured by overall survival (OS) | 2 years
  Overall survival (OS) will be determined as the time from the start of treatment until death due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of medical Oncology A450B Starling Loving Hall, Ohio City, Ohio, United States